CLINICAL TRIAL: NCT03783624
Title: A Randomized-controlled Clinical Trial of Hypnosis Versus Open Label Placebo for Chronic Neuropathic Pain With an Investigation of Neuro-cognitive Dysfunctions as Maintaining Factors and Therapeutic Targets
Brief Title: Measuring the Effects of Complementary Therapies in Chronic Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chantal Berna (Other)
Responsible Party: Sponsor-Investigator, Chantal Berna, Principal investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER-VD 2017- 00924
Record Dates: First submitted 2018-07-10; First posted 2018-12-21 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Neuropathic Pain
Keywords: hypnosis; open label placebo; neurocognitive measures; stress; induced pain; HRV
MeSH Terms: conditions — Neuralgia | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: due to the nature of the treatment (Open label placebo, hypnosis)patients and care providers will be in an open label setting, however the investigators and outcomes assessors will be blinded to the conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis (Experimental): This represents 6 individual script-based sessions lasting 1h, distributed over 8 weeks, administered by a certified expert in therapeutic hypnosis. A set of standardized recordings are provided to use at home for self-hypnosis. Suggestions address deep relaxation, sensory substitution or transformation, pain intensity reduction, decreased pain unpleasantness and intensity, sense of control. A brief example of such suggestions: "in this deeply relaxed state, you can imagine that your feet are covered in anesthetic… a deep layer of a powerful anesthetic medication, creating protective, soothing socks with which you can walk again…".
  Interventions: Behavioral: Hypnosis
- Open Label placebo (Placebo Comparator): This consists in information provided with a placebo pill. Patients are asked to take the placebo pills as a self-healing ritual. The information relies on 4 points of explanation, i.e. (1) the placebo effect can be powerful, (2) the body automatically can respond to taking placebo pills like Pavlov dogs who salivated when they heard a bell, (3) a positive attitude can be helpful but is not necessary, and (4) taking the pills faithfully for the full duration of treatment is critical.
  Interventions: Behavioral: Open label placebo
- Usual care (No Intervention): Patients continue with their usual treatments

INTERVENTIONS:
Behavioral: Hypnosis — A 6 session course of individual hypnosis therapy will be offered.
  Arms: Hypnosis
Behavioral: Open label placebo — Ritual intake of 2 placebo capsules twice a day
  Arms: Open Label placebo

SUMMARY:
The objective of the study is to a) assess the presence of a maladaptive stress response, a decreased pain modulation and any cognitive impairment in patients with chronic neuropathic pain in comparison to healthy controls. and b) evaluate the efficacy of a treatment of hypnosis and of an open label placebo on these neuro-cognitive factors and on clinical pain.

This will be done through a) a prospective observational comparative study of patients (base line measures) with Healthy Controls (HC) and b) an Open label; randomised, hypnosis vs. open label placebo (OLP) vs. treatment as usual control design; with a second phase of exploratory cross-over.

DETAILED DESCRIPTION:
The current study, through two sub-studies, aims to investigate through clinical, psychophysical and biological methodology in a population of patients with chronic neuropathic pain (i.e. involving a peripheral or CNS lesion), A) signs of a maladaptive stress response, correlates of decreased pain modulation, and of cognitive impairment, B) test hypnosis vs. open label placebo as potential mechanistic treatments of these suspected maintaining factors.

Patients will be recruited at the CHUV's Pain Center and via collaborating physicians treating patients with neuropathic pain (general practitioner, neurologist…). Controls will be recruited via advertisements posted in public places such as the CHUV, or the University of Lausanne's website and compounds.

Participants will be informed, in a clear and comprehensible way, of the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail.

Participants (patients and volunteers) will be first phone or live pre-screened by the study team to ensure they fulfil the inclusion criteria (except the MMSE). Then, eligible participants will be invited to the pain centre for the first study visit. During this visit informed will first be collected by the PI. Following this, a screening of the cognitive function of the participant will be performed through the MMSE test. Participants with a score lower than 24/30 will be excluded and informed of their exclusion and its cause. Pre-screening and/or screening data of non-included participants will be archived anonymously at the pain center in order to document the CONSORT diagram. All other consented participants will then take part in the first study procedures, which consist in a psychophysical assessment to determine their baseline performance. These will be compared between patients and matched volunteers without chronic pain, as well as longitudinally across treatment groups. This assessment lasts approximately 3h and includes physiological recording (cardiac rhythm, pulse-oxymetry, respiratory frequency), cognitive functions evaluation (Wisconsin cards sorting test, Trail Making Test, Complex Figure Copy) and questionnaires (Brief Pain Inventory, Hospital Anxiety and Depression Scale, Tampa Scale of Kinesiophobia, Pain Catastrophizing Scale, WHO-BREF quality of Life, Brief Resilience Scale, Pain coping, scale and sleep index). During this visit, patients will also undergo sensory testing to evaluate their abilities to modulate pain perception. Moderately painful 10s.heat stimuli will be applied on the forearm with a thermode (Medoc TSA, Israel). In pseudo-random order, participants are instructed to pay attention to the stimulus, vs. use distraction or focused mental imagery (i.e. reappraisal of the sensation). A peripheral blood plasma sample will also be collected for metabolomic analysis, in collaboration with the Metabolomics platform of the University of Lausanne. The day before the psychophysical assessment, participants will receive instructions for saliva collection in order to determine the variation of cortisol levels during the day (4 time points) and metabolomic signature. They will receive kits either directly or by mail. Participants will bring the samples along with them to the study visit.

Healthy volunteers will only participate in this unique visit. Patients will be randomized in equal proportions into the "Hypnosis", "Open Label Placebo" or the "treatment as usual" arm.

After 4 weeks, brief questionnaires will be filled regarding pain levels. After 8 weeks, all the patients will participate in the same psychophysical assessment as described above. Patients will also participate in the assessment of their hypnotisability. Afterward, we will proceed with an exploratory, patient-choice cross-over i.e. patients randomized in the "standard of care" arm will choose between the "hypnosis" or "open label placebo" arm. Those that initially received hypnosis treatment will be free to practice self hypnosis as taught during the treatment sessions, or switch to "open label placebo". Those in the "open label placebo" can choose to continue OLP or switch to hypnosis. All participants can also choose no further intervention.

After 16 and 24 weeks a follow-up questionnaire will evaluate the longer-term efficacy of the intervention and its impact on daily life, as well as adherence to treatment and satisfaction. Questionnaires will be filled online, from home.

The intervention consists in

1. . Hypnosis. This represents 6 individual script-based sessions lasting 1h, distributed over 8 weeks, administered by a certified expert in therapeutic hypnosis. A set of standardized recordings are provided to use at home for self-hypnosis. Suggestions address deep relaxation, sensory substitution or transformation, pain intensity reduction, decreased pain unpleasantness and intensity, sense of control. A brief example of such suggestions: "in this deeply relaxed state, you can imagine that your feet are covered in anesthetic… a deep layer of a powerful anesthetic medication, creating protective, soothing socks with which you can walk again…".
2. . Open label placebo. This consists in information provided with a placebo pill. Patients are asked to take the placebo pills as a self-healing ritual. The information relies on 4 points of explanation, i.e. (1) the placebo effect can be powerful, (2) the body automatically can respond to taking placebo pills like Pavlov dogs who salivated when they heard a bell, (3) a positive attitude can be helpful but is not necessary, and (4) taking the pills faithfully for the full duration of treatment is critical.

The active treatments are compared treatment as usual. Treatment as usual involves medications, interventional pain therapy, physical therapy, and psychotherapy as needed, provided by the patient's current physicians. Patients are required to be on stable medication 1 month prior to enrollment, and have no novel medication or procedures introduced during the 2 first months of the trial.

ELIGIBILITY:
Patients:

Inclusion criteria:

* aged 18-90 years,
* interested in complementary medicine
* peripheral neuropathic pain lasting for more than 6 months,
* pain intensity of at least 3/10 VAS over the last two weeks

Exclusion criteria:

* cognitive deficit (MMSE<24/30),
* severe hearing impairment,
* acute psychiatric (e.g. suicidality, psychotic symptoms) or somatic (e.g. unstable cardiorespiratory condition) co-morbidity preventing full engagement in the 8-week study intervention,
* prior negative experience with hypnosis,
* allergy or intolerance to mannitol.

Healthy controls:

Inclusion Criteria:

* matching patients for age and gender,
* no chronic pain condition no acute pain condition requiring daily intake of analgesics,
* no acute medical or psychiatric condition.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Interference due to pain (BPI interference) | at 8 weeks
  Brief Pain Inventory, mean interference with function score (score 0-10), with higher scores meaning higher interference.
pain severity (BPI pain scale) | at 8 weeks
  Brief Pain Inventory, mean pain intensity score over last 2 weeks (score 0-10) with higher scores meaning higher pain
fMRI of pain regulating circuitry (BOLD signal changes) | 8 weeks
  BOLD signal will be measured during pain perception

SECONDARY OUTCOMES:
Stress response measured through Cortisol awakening response | at 8 weeks
  Four sequential salivary samples at awakening will be collected and allow dosing of salivary cortisol levels (Cortisol Awakening Response curve).
Stress response measured through Heart rate variability (HRV) | at 8 weeks
  ECG collection over times of rest and induced stress will allow to calculate HRV (based mainly on the RR interval)
Pain modulation: modulation of induced pain through mental imagery and expectations. The outcome measure is on pain Visual Analogue Scale (VAS) for unpleasantness | at 8 weeks
  induced heat pain will be modulated through different instructions provided with visual cues: e.g. participants will be asked to imagine the stimulus is delivered in different contexts (more or less pleasant). The responses are given on a Pain unpleasantness Visual analogue Scale (VAS) ranging from 0 (not at all unpleasant: better outcome) to 10 (as much as can be unpleasant: worse outcome).
Pain modulation: modulation of induced pain through mental imagery and expectations. The outcome measure is on pain Visual Analogue Scale (VAS) for intensity | at 8 weeks
  induced heat pain will be modulated through different instructions provided with visual cues: e.g. participants will be asked to imagine the stimulus is delivered in different contexts (more or less pleasant). The responses are given on a Pain intensity Visual analogue Scale (VAS) ranging from 0 (not at all intense- better outcome) to 10 (as much as can be intense- worse outcome).
Trail making test (outcomes in time, seconds) | at 8 weeks
  Neuro-cognitive functioning testing
Wisconsin card sorting task | at 8 weeks
  Standardized cognitive flexibility task
Rey-Osterrieth figure test | at 8 weeks
  Prospective thinking task
Hospital Anxiety and Depression Scale (HADS) | at 8 weeks
  Hospital Anxiety and Depression Scale (HADS), which measures anxiety and depression symptoms in patients with somatic medical diagnosis. This scale ranges from 0-42 points, where higher scores indicate more depression/Anxiety. There are 2 sub-scales, each with 21 points, one for depression, teh other one for anxiety. The global scale score is calculated as a total
Tampa Scale of Kinesiophobia | at 8 weeks
  Tampa scale of fear of movement (i.e. Kinesiophobia): A scale with results ranging from 11-44 points, with teh higher points suggesting more severe kinesiophobia (worse fear of movement, worse outcome).
Pain Catastrophizing Scale (PCS) | at 8 weeks
  This scale measures the Catastrophizing thinking regarding pain scale. The score ranges between 0-52 with the higher scores indicating more severe catastrophizing, i.e. worse negative thinking regarding pain.
Coping Strategies Questionnaire | at 8 weeks
  Scale measuring the cognitive coping strategies used to deal with pain, with scores ranging from 0 to 78 points total, with higher scores indicating higher coping skills
patient satisfaction with care | 4 and 8 weeks
  Subjective measure of satisfaction with the treatment, on a VAS scale: How satisfied are you with your attributed treatment? VAS 0: not at all; 10: very much satisfied
Evaluation of patient compliance | 4 and 8 weeks
  Subjective measures of compliance: adequate adherence to treatment recommendations: question : "were you able to follow the treatment plan as instructed? " Yes/no" if no: why. NUmber of patients reporting adequate compliance.
Blood metabolomics | 8 weeks
  Metabolomics is the analysis of the metabolic state (metabolites in the blood, saliva or other bodily fluid) at a given time. It is a growing technology that allows to analyse the biological response from a broader perspective and offers a sensitive way to investigate poorly-explored biochemical pathways in disease. The analysis of metabolites may provide a technically and bioinformatically tractable, physiologically relevant, chemically comprehensive method to better understand complex chronic diseases. For example, a recent study on chronic fatigue syndrome (CFS) showed an objectively identifiable chemical signature in both men and women with CFS distinct from healthy controls. Metabolomics showed that CFS is a highly concerted hypometabolic response to environmental stress that traces to the mitochondria.

OTHER OUTCOMES:
second phase cross-over choice | 8 weeks
  patients are offered to choose a second treatment at 8 weeks
Long term outcomes on the Brief Pain Inventory (BPI) | 24 weeks
  brief pain inventory, which measures the average pain score (pain VAS 0: no pain to 10: worst pain, and pain interference = no interference on daily activities by pain, 10 = full interference (see outcomes 1-2)
expectations regarding treatment effects | 8 weeks, 24 weeks
  measured at Baseline: Question: how well do you expect this treatment to work for you (VAS: 0: no effect at all to 10: full relief).
Hypnotisability according to the Carleton University Responsiveness to Suggestion Scale (CURSS) | 8 weeks
  This scale The Carleton scale yields 3 suggestibility scores for each S: objective (CURSS-O) scores reflect overt response to suggestion, subjective scores reflect experiential response to suggestion. Objective scores range from 0-7 , subjective scores from 0-21. The higher the score, the more hypnotizable the people are.

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital (CHUV), Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data can be made accessible to interested researchers upon request